CLINICAL TRIAL: NCT01453140
Title: Phase I- II Study of in Vivo Regulatory T Cell Enhancement With Cyclophosphamide and Sirolimus With or Without Vidaza (Azacitidine) for the Treatment of Steroid-refractory Acute Graft-versus-host Disease
Brief Title: In-vivo Regulatory T Cell Enhancement With Cyclophosphamide and Sirolimus
Acronym: T-REG
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Dose Limiting Toxicities
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREG - Pro2219
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; Sirolimus; Interleukin-2; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cyclophosphamide and Sirolimus (Experimental): cyclophosphamide and sirolimus combo
  Interventions: Drug: Cyclophosphamide and Sirolimus
- Lowdose IL-2, Cytoxan + Sirolimus (Experimental): Low dose IL-2 with Cytoxan + Sirolimus Patients in treatment arm B will be receiving low-dose IL-2 in conjunction with the cyclophosphamide and sirolimus.
  Interventions: Drug: Low dose IL-2 with Cytoxan + Sirolimus
- Lowdose IL-2, Vidaza, cyclophosphamide & Sirolimus (Experimental): Lowdose IL-2, Vidaza, cyclophosphamide (Cytoxan) & Sirolimus Patients in treatment arm C will be receiving low-dose azacitidine (Vidaza).
  Interventions: Drug: Low dose IL-2, low dose Vidaza, cyclophosphamide & Sirolimus; Drug: Low dose IL-2, Vidaza, Cytoxan & Sirolimus

INTERVENTIONS:
Drug: Cyclophosphamide and Sirolimus — On the first day of treatment, cyclophosphamide will be administered at a dose of 4g/m2 IV x 1 dose. Patients who are >40% above ideal weight will be dosed based on adjusted weight and adjusted BSA.
  One day after the administration of cyclophosphamide, patients will receive sirolimus 6 mg PO x 1 and on the following day will start sirolimus at a dose of 2 mg PO daily.
  Other Names: Cytoxan
  Arms: Cyclophosphamide and Sirolimus
Drug: Low dose IL-2 with Cytoxan + Sirolimus — Patients in treatment arm B will be receiving low-dose IL-2 in conjunction with the cyclophosphamide and sirolimus.
  IL-2 will be administered at a dose of 0.5E6 IU/m2 SQ daily x 8 weeks followed by 4 weeks off, starting 14 days after the cyclophosphamide.
  Other Names: Interleukin-2; Cytoxan
  Arms: Lowdose IL-2, Cytoxan + Sirolimus
Drug: Low dose IL-2, low dose Vidaza, cyclophosphamide & Sirolimus — Patients in treatment arm C will be receiving low-dose azacitidine (Vidaza). The Vidaza will be initiated between day 27 and 32 following the cyclophosphamide.
  The dose administered will be 10 mg SQ daily for 5 days followed by 3 weeks off.
  Other Names: Interleukin-2; Azactidine; Cytoxan
  Arms: Lowdose IL-2, Vidaza, cyclophosphamide & Sirolimus
Drug: Cyclophosphamide and Sirolimus — Day 1: Cyclophosphamide Day 2: Sirolimus
  Other Names: Other names: Cytoxan
  Arms: Cyclophosphamide and Sirolimus
Drug: Low dose IL-2 with Cytoxan + Sirolimus — treatment arm B will be receiving low-dose IL-2 in conjunction with the cyclophosphamide and sirolimus
  Other Names: Other names:; Interleukin-2; Cytoxan
  Arms: Lowdose IL-2, Cytoxan + Sirolimus
Drug: Low dose IL-2, Vidaza, Cytoxan & Sirolimus — Vidaza will be initiated between day 27 and 32 following the cyclophosphamide.
  Other Names: Other names:; Interleukin-2; Azactidine; Cytoxan
  Arms: Lowdose IL-2, Vidaza, cyclophosphamide & Sirolimus

SUMMARY:
In this study the investigators are proposing to treat patients with steroid-refractory Graft-versus-host Disease (GVHD) stabilization using IL-2 and azacitidine

DETAILED DESCRIPTION:
High-dose cyclophosphamide and sirolimus have been successfully used for the prevention of Graft-versus-host Disease (GVHD) and have shown to enhance the Tregs subpopulation. The addition of low dose IL-2 and a demethylating agent such as azacitidine will also be studied in an attempt to promote and stabilize the FoxP3 expression of Tregs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented clinical diagnosis of grade II-IV acute graft-versus- host disease defined as graft versus host disease (GVHD) occurring within the first 100 days of transplantation
* Patients must be steroid-refractory defines as progression after 3 days of corticosteroid therapy or no response after 5 days of corticosteroid therapy.
* Progression is defined as up-grading
* No response is defined as no down-grading
* Progression after 3 days requires patients to have received at least 2 mg/mg/day for a total of 6 mg/kg of methylprednisolone or its equivalent.
* No response after 5 days requires patient to have received at least 2 mg/kg/d for a total of 10 mg/kg of methylprednisolone or its equivalent.
* Patients with exacerbation of GVHD during steroid taper will require re-treatment with 2mg/kg/d of corticosteroids and will need to meet the criteria
* Age 18-70
* Patients must have received an allogeneic hematopoietic stem cell transplant within 100 days of study enrollment.
* Serum creatinine < 2 mg/dL

Exclusion Criteria:

* Patients cannot have active central nervous system (CNS) disease.
* Patients must not have received cyclophosphamide for GVHD prophylaxis
* Patients must not have pneumonia requiring oxygen supplementation
* Unable or unwilling to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4/11/2011 - 5/1/2013 - recruitment at Hackensack University Medical Center
Pre-assignment Details: Pts.must have a documented clinical diagnosis of grade II-IV acute graft-versus- host disease defined as GVHD (graft versus host disease) within 100 days p transplantation.
  Patients must be steroid-refractory defined as progression after 3 days of corticosteroid therapy or no response after 5 days of same. see study details.
Groups:
- Cyclophosphamide and Sirolimus Only: Cyclophosphamide = 4g/m2 IV Sirolimus = 6 mg PO x 1; 2 mg PO
  No patients were enrolled in the Cyclophosphamide, Sirolimus, IL-2 arm or the Cyclophosphamide, Sirolimus, IL-2, azacitidine arm
Period: Overall Study
Arm/Group | Cyclophosphamide and Sirolimus Only
Started | 3 (3 patients were enrolled)
Completed | 0 (All three patients experienced grade 4 limiting toxicities (possible treatment related))
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Three subjects started the study - all three had limiting toxicities and died. Study was terminated
Groups:
- Cyclophosphamide and Sirolimus: Patients will be treated in sequential cohorts of 5. In cohort A, the first 5 enrolled patients will be receive cyclophosphamide and sirolimus only
Arm/Group | Cyclophosphamide and Sirolimus
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — number of subjects in age categories
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 1
    Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Patients With Steroid-refractory Graft-versus-host Disease (GVHD) Using Cyclophospahmide and Sirolimus Combined With 3 Variations of Low-dose IL 2 and Low-dose Vidaza.
Description: The primary objective of this study is to determine the response rate of patients treated steroid-refractory graft-versus-host disease (GVHD) using cyclophospahmide and sirolimus combined with 3 variations of low-dose IL 2 and low-dose Vidaza with an outcome goal of promoting CD4+CD25+FoxP3+ Tregs.
Time Frame: 28 days to 100 days post transplant
Population: No patients were enrolled in the Low dose IL-2 with Cytoxan + Sirolimus or Low dose IL-2, Vidaza, Cytoxan & Sirolimus arms
Measure: Number; unit: Participants
Groups:
- Low Dose IL-2 With Cytoxan + Sirolimus: Patients in treatment arm B will be receiving low-dose IL-2 in conjunction with the cyclophosphamide and sirolimus.
- Low Dose IL-2, Vidaza, Cytoxan & Sirolimus: Patients in treatment arm C will be receiving low-dose azacitidine (Vidaza)
Arm/Group | Cyclophosphamide and Sirolimus | Low Dose IL-2 With Cytoxan + Sirolimus | Low Dose IL-2, Vidaza, Cytoxan & Sirolimus
Number analyzed (Participants) | 3 | 0 | 0
Participants | 0 |  |

ADVERSE EVENTS:
Time Frame: SAE data was collected over a period of 6 months for the three patients enrolled in the study
Description: Please see SAE # 5045 and 5063 SAE # 5633 and 5878 and SAE 5055 for h/o DVT, CMV+ -dated 10-18-11 SAE 5247 for diarrhea and fever - dated 12-13-11 SAE 5379 for severe anemia dated 1-10-12 SAE 5899 for new brain masses vs abscess dated 4-6-12 SAE 5917 for confusion,malaise weakness dated 4-23-12
Groups:
- Cyclophosphamide and Sirolimus: Cyclophosphamide and Sirolimus - Patients will be treated in sequential cohorts of 5. In cohort A, the first 5 enrolled patients will be receive cyclophosphamide and sirolimus only
- Low Dose IL-2 With Cytoxan + Sirolimus: Low dose IL-2 with Cyclophosphamide + Sirolimus - In cohort B, the next 5 patients will additionally receive cyclophosphamide and sirolimus & low-dose IL-2 Low dose IL-2, low dose Vidaza, Cyclophosphamide & Sirolimus
- Low Dose IL-2, Vidaza, Cytoxan & Sirolimus: Low dose IL-2, Vidaza, Cytoxan & Sirolimus - In cohort C the next 5 enrolled patients will additionally receive cyclophosphamide and Sirolimus, low-dose IL-2 and low-dose Vidaza
Arm/Group | Cyclophosphamide and Sirolimus | Low Dose IL-2 With Cytoxan + Sirolimus | Low Dose IL-2, Vidaza, Cytoxan & Sirolimus
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide and Sirolimus (N=3) | Low Dose IL-2 With Cytoxan + Sirolimus (N=0) | Low Dose IL-2, Vidaza, Cytoxan & Sirolimus (N=0)
SAE 5379 - Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — 5379-1/10-2012- Blood test revealed anemia, rated as category 3 severe, affecting subject 1, possibly treatment related
SAE 5917-neurological (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — 5917 - 4/23/2012 - Upon examination using scans based on symptoms, pt 1 was found to have neurological symptoms related to transplant hospitalized, and categorized as serious - rated 3
SAE 6031- Post-transplant lymphoproliferative disorder (PTLD) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — 6031- 5/22/2012 - Pt developed post transplant lymphoproliferative disorder due to GVHD reseulting in death, rated as severe
SAE 5063 - C. difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — 5063- 10-22-2011 - Pt 2 experienced severe refractory GVHD and c diff infection resulting in death on 10-22-2011, listed as severe - category 5, and possibley related to treatment
SAE 5878- Graft Versus Host Disease (GVHD) (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — 5878 - 4/15/2012 - Pt 3 experienced severe grade 4 GVHD of liver resulting in death, rated as severe, category 5 and possibly related to condition/treatment
SAE 5856-brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — 5856- 4/6/2012 - Pt 1 experienced new brain masses found on cat scan and erythema around rt eye, rated as category 3, Serious and listed as a known possible side effect of treatment
SAE 5055- Deep vein thrombosis (DVT) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — 5055- 10-13-2011 - Pt 1 admitted to hospital for treatment of new brain tumor or abcess, rated as category 2, and category 3, and listed as known side effect of transplant chemo
Deep Vein Thrombosis, Cytomegalovirus infection and Graft Versus Host Disease Complications (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Pt 1 was admitted for treatment of left upper extremity DVT, CMV infection and GVHD complications - categorized as serious level 3 and listed as possible treatment related

LIMITATIONS AND CAVEATS:
3 patients enrolled - all 3 had grade 4 (possibly treatment related) limiting toxicities. All three patients have since passed away. Study was closed after being on hold as per stopping rules.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes